CLINICAL TRIAL: NCT03327441
Title: Benefits of Almond Consumption in Modulation of Intestinal Microbiome and Novel Disease Risk Biomarkers: A Randomized Controlled Dietary Intervention Trial
Brief Title: Benefits of Almond Consumption in Modulation of Intestinal Microbiome and Novel Disease Risk Biomarkers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of the funder: Almond Board of California
Sponsor: University of Manitoba (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B2017:105
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2021-04

CONDITIONS: Microbiota
MeSH Terms: interventions — Rab1 protein, Drosophila

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonds (Experimental)
  Interventions: Other: Almonds
- Omelette (Active Comparator)
  Interventions: Other: Omelette

INTERVENTIONS:
Other: Almonds — Almonds will be provided as 15% energy
  Arms: Almonds
Other: Omelette — Omelettes will be provided as 15% energy
  Arms: Omelette

SUMMARY:
The overall goal is to assess the health benefits of almond consumption on gut microbiome patterns and their association with circulating disease risk biomarkers, as well as the processes that control those pathways. Health benefits will be assessed relative to a omelette control.

DETAILED DESCRIPTION:
Men and women with elevated waist circumference aged between 18-75 yrs will be recruited from the Winnipeg (Manitoba, Canada) area to participate in a two arm crossover, randomized study; each treatment period will be 4 weeks in length, with a 4 week washout period separating each treatment. Participants will be randomized to consume either i) almonds, or ii) omelettes at 15% of energy. Each of the treatment products will contain equal levels of calories.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* Men and women 18-75 yr
* Elevated waist circumferences (women greater than or equal to 80 cm, men greater than or equal to 94 cm)
* LDL-C greater than or equal to 2.8 mmol/L, or less than or equal to 4.9 mmol/L
* Non-smokers
* Possess a telephone or email address to enable regular contact
* Able to read, write and speak English

Exclusion Criteria:

* Pregnant female, or planning to become pregnant during the study period
* Weight gain or loss of at least 10lbs in previous three months
* Allergic to almonds, eggs, milk
* Exercising > 15 miles/wk or 4,000 kcal/wk
* Those currently taking (or have taken within the past 3 months) lipid-lowering medications (i.e., statins)
* Those currently taking (or have taken within the last 3 months) lipid-lowering supplements (i.e., omega-3 supplements, plant sterols/stanol foods and/or supplements, fibre, etc.)
* Those currently taking (or have taken within the last 3 months) probiotic supplements and foods containing added probiotics (i.e., kefir, Activia, Kashi: Vive Probiotic Digestive Wellness Cereal)
* Previous history of diabetes, hypertension, gastrointestinal disease, liver or lung disease or cancer, hyperthyroidism or hypothyroidism, or lung disease.
* Alcohol use of >2 drinks/day

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal microbiome | 4 weeks
  Bacterial community alpha-diversity measured using richness and diversity indices including Chao1, Shannon, Inverse Simpson.
  Bacterial community beta-diversity measured using weighted and unweighted UniFrac distances.
  The most abundant Operational Taxonomic Units (OTUs) within the bacterial community identified based on the relative abundances of the OTUs within the community.
  Bacterial community composition at the phylum and genus levels described based on the relative abundances of each taxa within the community.
  Bacterial community functional capacity measured based on the relative abundances of collected predicted functions of the community members.
  Ecological relationships between members of bacterial community assessed using correlation network modelling to identify keystone and foundation members of the bacterial community that have the highest number of positive (supportive) or negative (suppressive) connections (>15) with other members of community.

SECONDARY OUTCOMES:
Blood total cholesterol | 4 weeks
Blood low-density lipoprotein cholesterol | 4 weeks
Blood high-density lipoprotein cholesterol | 4 weeks
Blood triglycerides | 4 weeks
Interferon gamma | 4 weeks
Interleukin 1 beta | 4 weeks
Interleukin 6 | 4 weeks
Tumor necrosis factor alpha | 4 weeks
Serum amyloid A | 4 weeks
C-reactive protein | 4 weeks
Vascular cell adhesion molecule 1 | 4 weeks
Intercellular adhesion molecule 1 | 4 weeks
7α-hydroxy-4-cholesten-3-one | 4 weeks
Fecal short chain fatty acids | 4 weeks
Fatty acid synthesis rate | 4 weeks
Cholesterol synthesis rate | 4 weeks
Cholesterol absorption rate | 4 weeks
Body mass index | 4 weeks
  Weight and height will be combined to report BMI in kg/m^2
Waist circumference | 4 weeks
Hip circumference | 4 weeks
Blood pressure | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rotimi Aluko, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada